CLINICAL TRIAL: NCT00522613
Title: Recovery Group Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Portland State University (Other); University of South Florida (Other)
Responsible Party: Stanley Watson, Kaiser Foundation Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NW-05CGREE-01
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2006-09

CONDITIONS: Bipolar Disorder; Schizophrenia; Schizoaffective Disorder
Keywords: recovery; serious mental illness; bipolar disorder; schizophrenia; schizoaffective disorder
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Recovery Group Project — Recovery Group Workbook & Group Sessions

SUMMARY:
The purpose of this study is to develop and evaluate a low-cost, joint consumer/counselor-led, health education and support intervention that will foster self-care and recovery among adults with serious mental illness. Results from the study will indicate how well the workbook and the overall program were received by individuals with serious mental illness, and whether participating in the program appeared to improve recovery and functioning.

DETAILED DESCRIPTION:
Recent research suggests that many individuals with serious mental illnesses may recover from these conditions and become fully integrated into their communities. Although improved medications may be most responsible for these developments, self-help groups, social support, and empowerment have been identified as important facilitators of the recovery process. Recovery-oriented, consumer-led approaches are gaining in popularity, but few of these interventions have been evaluated scientifically.

This pilot study proposes to develop and evaluate a recovery-oriented program that centers on the use of a self-help workbook. Results from the study will indicate how well the workbook and the overall program were received by individuals with serious mental illness, and whether participating in the program appeared to improve recovery and functioning.

Objectives:

1. To develop group-facilitator materials to complement the self-help workbook.
2. To conduct a randomized trial of the intervention with kaiser Permanente Northwest (KPNW) members with bipolar disorder or schizophrenia/schizoaffective disorder, using a delayed control group design and 6- and 12-month post-intervention follow-up.
3. To assess participant attendance and satisfaction with the group sessions;
4. To assess whether participating in the group intervention was associated with improvements in short-term recovery and functioning.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bipolar disorder or schizophrenia/schizoaffective disorder
* current membership in KPNW
* age 18 or over

Exclusion Criteria:

* having a guardian
* psychotic symptoms that interfere with group interactions
* dementia, mental retardation (other than mild) or other organic brain conditions that affect an individual's ability to participate in an interview, a group intervention, or complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To develop group-facilitator materials to complement the self-help workbook | 6 weeks
To conduct a randomized trial of the intervention with KPNW members | 6 weeks
To assess participant attendance and satisfaction with the group sessions | 6 weeks
To assess whether participating in the group intervention was associated with improvements in short-term recovery and functioning | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carla A. Green, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States